CLINICAL TRIAL: NCT06990789
Title: Effect of Self-Applied Ear Massage on Sleep Quality of Earthquake-Affected Women
Brief Title: Ear Massage and Sleep Quality in Earthquake-Affected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Demet Harbalioğlu, Master's student, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinU-SBE-DH-01
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Sleep Quality; Sleep Perception
Keywords: sleep; woman; ear massage; Earthquake
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: two groups with a self-ear massage control group
Who Masked: Participant
Masking Description: The women participating in the study will not know which group they belong to. During the statistical analysis of the study, group codes will be designated as A and B, and which code represents which group will be kept in a sealed envelope by a researcher who is not involved in the analysis process. Once all analyses are completed, the group codes will be revealed, thereby enhancing the impartiality and reliability of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group ear massage (effective ear massage) (Active Comparator): self ear massage will be applied to individuals starting from the endocrine point and occiput point located in the frontal lobe of the ear, massage is done to the heart, shenmen and sympathy points.
  Interventions: Behavioral: effective self-applied ear massage
- Control (Sham) Group Ear Massage (Sham Comparator): It will be applied to the five points called helix 1,2,3,4,5 located on the auricle. Care will be taken not to create pressure and a stroking movement will be made.
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: effective self-applied ear massage — The women will be treated for two weeks. It will be applied 7 days a week, in the first hour after waking up in the morning and in the last hour before going to bed at night. Each session will be 3 minutes.
  Arms: Intervention group ear massage (effective ear massage)
Behavioral: Sham Comparator — The women will be treated for two weeks. It will be applied 7 days a week, in the first hour after waking up in the morning and in the last hour before going to bed at night. Each session will be 3 minutes.
  Arms: Control (Sham) Group Ear Massage

SUMMARY:
The purpose is study is to vestigate the effect of self-administered ear massage on the sleep quality of women affected by the earthquake.

DETAILED DESCRIPTION:
Sleep is a necessary process for the body to renew and maintain functions. Sleep, which begins with the activation of the anterior hypothalamus region in the brain, occurs in two main stages: REM (Rapid Eye Movement) and NREM (Non-Rapid Eye Movement). The REM stage is associated with cognitive functions and memory, while the NREM stage supports cellular renewal and growth. While growth hormone and melatonin increase during sleep, cortisol levels decrease and the body prepares for the new day.

Sleep has a great role in regulating mental and physical health. However, sleep disorders are common in society and are seen in 22-50%. These disorders can lead to serious consequences such as concentration and memory problems, depression, immune weakness, obesity and heart diseases. Traumatic events such as earthquakes in particular trigger sleep problems and negatively affect the quality of life of individuals. Sleep disorders can continue for many years in people affected by earthquakes, and women are at higher risk in this regard.Socioeconomic conditions and psychiatric sensitivity in women contribute to the increased risk of sleep disorders.

Pharmacological and non-pharmacological treatments are used together to eliminate sleep disorders. While pharmacological methods can cause side effects, nonpharmacological approaches are safe and widely preferred. Ear massage, one of the nonpharmacological methods, is an effective intervention that can be applied independently in nursing care. The ear contains an important branch of the vagus nerve, and massage applied to this area activates the parasympathetic nervous system, contributing to stress reduction, balancing cortisol levels, and increasing sleep quality.

Ear massage stands out as an effective and side-effect-free method for individuals experiencing sleep problems after a disaster. It is of critical importance for public health nurses to develop and disseminate such easily applicable approaches, especially in the post-disaster period. Ear massage, which supports general health by stimulating the vagus nerve, offers an important option for improving individuals' sleep patterns and quality of life after traumatic events.

ELIGIBILITY:
Inclusion Criteria:

* Those with a PSQI score above 5 Women between the ages of 18-65 Those who volunteered to participate in the research and signed an informed form Those residing in Hatay during the earthquake Those who understand Turkish speech Those who have no obstacles to communication

Exclusion Criteria:

* Those who do not volunteer to participate in the study Those who experience chronic pain of unknown cause Those who have a disease diagnosed by a doctor (obstructive sleep disorder, psychiatric disorders, dementia, Alzheimer's disease, etc., cancer) Those who are pregnant or suspected of being pregnant Those who use prescription/non-prescription medications for sleep

  * Those who are receiving ongoing complementary therapy (e.g. aroma therapy, massage therapy, foot reflexology, yoga and tai chi)
  * Those who use food supplements/teas for sleep
  * Those with auricular plasia or hypoplasia
  * Those who have an active infection or skin integrity disorder in the ear area (ulcer, eczema, urticaria, surgical incision, etc.)
  * Those who have responsibilities such as taking care of a baby or the elderly that require waking up at night
  * Those who work shift jobs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 60 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
PSQI | Pre-test phase and 4 weeks after the post-test
  PSQI is a 19-item questionnaire to measure sleep quality, with a total score ranging from 0 to 21; lower scores indicate better sleep quality.
Xiaomi Smart Band 9 | 4 weeks (Pre-test phase, intervention phase, and post-test phase)
  It is planned to objectively measure sleep quality using the Xiaomi Smart Band 9 device. Xiaomi Smart Band 9, a small and portable device usually worn on the wrist, provides information about sleep-wake cycles by recording the user's movements. The data collected includes information such as sleep duration, time to fall asleep, night wakings, etc. Thus, objective and reliable data are obtained about individuals' sleep quality, daily activity levels and sleep patterns.
pre-sleep arousal scale | Pre-test phase and 4 weeks after the post-test
  The scale, which was developed to assess cognitive and somatic arousal levels in the pre-sleep phase, consists of 16 items and has two sub-dimensions assessing cognitive and somatic arousal before sleep. The items are rated on a 5-point Likert-type scale ranging from 1 (not at all) to 5 (very much). High scores obtained from the scale indicate high arousal.
readiness assessment form | pre-test phase
  This form includes the ear massage steps and was prepared to evaluate whether the participants performed the ear massage as intended at the end of the training.
Massage Application Tracking Form | two weeks
  Participants are asked to indicate the date and time of their ear massage twice a day for 14 days and whether they applied it or not.

CONTACTS AND LOCATIONS:
Overall Officials: OVERALL STUDY OFFİCİALS sümbüle köksoy vayısoğlu, doçent doktor, Study Director — Mersin University
Locations (1):
- Abdulgani Turkmen Konteynerkent, Hatay, DEFNE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Temel, A. B. (2022). Sağlığı koruma ve geliştirmede uyku sağlığı ve uyku hijyeni. In A. B. Temel (Ed.), Sağlığı koruma ve geliştirme (ss. 94-98). Ankara: Ema Tıp Kitabevi.